CLINICAL TRIAL: NCT00001275
Title: Ovarian Follicle Function in Patients With Primary Ovarian Insufficiency
Brief Title: Ovarian Follicle Function in Patients With Primary Ovarian Failure
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910127; 91-CH-0127
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-02-08

CONDITIONS: Amenorrhea; Hypoaldosteronism; Hypogonadism; Infertility; Premature Ovarian Failure
Keywords: Menopause; Estrogen; Infertility; Ovulation; Amenorrhea; Hypergonadotropic Hypogonadism; Young Women; Gonadal Steroid Deficiency; Mineralocorticoid Deficiency; Premature Ovarian Failure; POF
MeSH Terms: conditions — Amenorrhea; Hypoaldosteronism; Hypogonadism; Infertility; Primary Ovarian Insufficiency; Adrenal Insufficiency

SUMMARY:
No proven therapy to restore ovarian function and fertility is available to patients with karyotypically normal spontaneous premature ovarian failure. We know that one-half of these patients have primordial follicles remaining in the ovary, and these follicles can function intermittently. This is a diagnostic omnibus protocol that permits baseline clinical evaluation of patients with prematurem ovarian failure. The findings will determine patients' suitability for specifically focused therapeutic research protocols.

DETAILED DESCRIPTION:
No proven therapy to restore ovarian function and fertility is available to patients with karyotypically normal spontaneous primary ovarian insufficiency. We know that more than one-half of these patients have primordial follicles remaining in the ovary, and these follicles can function intermittently. This protocol permitted baseline clinical evaluation of patients with primary ovarian insufficiency and ongoing observation of the natural history of the disorder. The protocol is now in the follow up and analysis phase and is not now recruiting new patients. Now a major aim of the protocol is to investigate large scale medical sequencing as a method by which to uncover mechanisms of primary ovarian insufficiency and to assist in the management of women with this condition. This will involve a community-based participatory research approach.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women 18 to 42 years of age with primary ovarian insufficiency who meet the following requirements were candidates for recruitment to the study: 1) at least a four month history of oligo-amenorrhea not due to pregnancy, and 2) clearly elevated gonadotropins in the menopausal range on two separate occasions at least one month apart.

EXCLUSION CRITERIA:

Women with evidence for karyotypic, metabolic, toxic, or iatrogenic cause of the ovarian insufficiency were not candidates.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1134 (Actual)
Dates: Start 1991-05-12; Study Completion 2017-02-08

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence M Nelson, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nelson LM, Anasti JN, Kimzey LM, Defensor RA, Lipetz KJ, White BJ, Shawker TH, Merino MJ. Development of luteinized graafian follicles in patients with karyotypically normal spontaneous premature ovarian failure. J Clin Endocrinol Metab. 1994 Nov;79(5):1470-5. doi: 10.1210/jcem.79.5.7962345.
- [Background] Anasti JN, Flack MR, Froehlich J, Nelson LM. The use of human recombinant gonadotropin receptors to search for immunoglobulin G-mediated premature ovarian failure. J Clin Endocrinol Metab. 1995 Mar;80(3):824-8. doi: 10.1210/jcem.80.3.7883837.
- [Background] Kim TJ, Anasti JN, Flack MR, Kimzey LM, Defensor RA, Nelson LM. Routine endocrine screening for patients with karyotypically normal spontaneous premature ovarian failure. Obstet Gynecol. 1997 May;89(5 Pt 1):777-9. doi: 10.1016/s0029-7844(97)00077-x. PMID 9166320